CLINICAL TRIAL: NCT04944823
Title: Characterization of Cellular Immunology, Biochemical and Lung Microbiome, Correlated With the Development of Ventilation Associated Pneumonia (VAP) in Adult Patients Admitted to the Intensive Care Unit (ICU): The Second Stage.
Brief Title: Characterization Immunology, Biochemical and Lung Microbiome, Correlated With the Ventilation Associated Pneumonia (VAP)
Acronym: MicroNAV-II
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Other Study IDs: MED-286-2020
Record Dates: First submitted 2021-06-10; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: pulmonary microbiome; SARS-CoV Infection; Covid19
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — orotracheal secretion Rectal swab bronchoalveolar lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID 19 infection who develop bacterial coinfection.: Follow-up for 24 months
  Interventions: Other: Clinical follow-up for 24 months
- Patients with COVID 19 infection who do not develop bacterial coinfection.: Follow-up for 24 months
  Interventions: Other: Clinical follow-up for 24 months

INTERVENTIONS:
Other: Clinical follow-up for 24 months — Sampling and clinical follow-up for 24 months

SUMMARY:
SARS-CoV-2, the virus that causes COVID-19, is currently a global public health problem, declared a pandemic by the World Health Organization, which today has more than one million deaths in the world, of which , 30,000 approximately belong to Colombia, being the country number 11 with the highest number of deaths. The most common symptoms related to this disease are fever, cough, dyspnea, myalgia, headache, diarrhea and rhinorrhea. COVID-19 is characterized by immune system dysfunction and hyperinflammation causing acute respiratory distress syndrome, macrophage activation, and coagulopathy. The clinical course for SARS-CoV-2 in most cases is mild, but approximately 14% of cases can be severe. In pneumonia caused by SARS-CoV-2, the lung lining is known to alter the composition of the lung microbiome, in addition to lymphocyte damage that can promote the growth of bacteria to initiate bacterial pneumonia, and it is estimated that the prevalence of coinfection / superinfection reaches 50% among deaths from COVID-19. Coinfection between different microorganisms and SARS-CoV-2 is a serious problem in the COVID-19 pandemic, and there is still little information on this.

It is for this reason that the researchs propose to develop this research project that will allow to understand the possible mechanisms associated with the development of bacterial coinfection / superinfection in patients diagnosed with COVID-19, which will allow expanding the panorama of knowledge towards a better and adequate treatment in these patients, as well as detection of biomarkers or clinical phenotypics that may be useful in the diagnosis, based on evidence.

It is important to note that these results are of clinical importance since we will try to identify biomarkers or changes in the lung microbiome that allow doctors to early identify patients at risk of developing coinfection and thus initiate early treatments or preventive measures, which allow the improvement of clinical outcomes in patients. Results will be presented in a timely manner at national and international conferences and in peer-reviewed, indexed, high-impact journals.

DETAILED DESCRIPTION:
This is a prospective, translational (T0-T2), multicenter, observational, cohort study of consecutive patients with a first clinical phase, where the collection of different types of samples (Bronco alveolar lavage, blood, nasopharyngeal swab, secretion orotracheal and rectal swabbing) at the start of mechanical ventilation, on day 3 and before extubation and another stage of molecular analysis in human samples collected where by different types of techniques such as: characterization of the 16S ribosomal unit, ELISA, time PCR real, concentration and cell discrimination techniques, we will characterize the microbiological, immunological and cellular changes that condition the development of coinfection.

Descriptive analytical studies, techniques, and parametric and nonparametric tests will be used to explore diagnostic, microbiological, or subgroup differences, as well as clinical outcomes. Independent predictors and associated hazard ratios with 95% confidence intervals will be reported. A two-tailed p value less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU, COVID-19 positive by RT-PCR, who require assisted mechanical ventilation.
* Adult patients over 18 years of age.
* Patients who agree to participate in the study and sign the informed consent form (family members or legal representative).
* Patients in whom the identification of the causative agent of coinfection is attempted within the first 48 hours of hospitalization.

Exclusion Criteria:

* Patient on mechanical ventilation for more than 24 hours without being evaluated for study entry.
* Patient who was treated with antibiotics 7 days prior to hospitalization or time of assessment for the study.
* Pregnant or breastfeeding patients.
* People who belong to population groups with increased vulnerability such as, for example, prison population, minors detained in orphanages or people in street situations.

No research procedure, clinical or paraclinical, or taking of clinical information or biological samples will be performed before the patient or his/her legal representative agrees to participate in the study and signs the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit of the Clínica Universitaria de la Sabana, with a diagnosis of COVID-19 by RT-PCR, who require invasive mechanical ventilation due to respiratory failure as a result of the infection and who approve their participation in the study. It is important to highlight that these patients are sedated and cannot agree to participate in the study; therefore, the patient's relatives or legal representative will be in charge of defining the participation of the relative in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Identification of the pulmonary microbiome and changes in microbial diversity in patients with severe COVID. | 24 months
  To observe the change that occur in the diversity of the pulmonary microbiome in patients with severe COVID, with mechanical ventilation. The pulmonary microbiome will be analyzed at 4 four times during the patient's mechanical ventilation (baseline, 72 hours, fifth day, seventh day or if he/she develops co-infection or superinfection).
Correlation between microbial diversity and host immune response with severe COVID. | 24 months
  To analyze whether changes in microbial diversity have any association with the host immune response leading to increased susceptibility to co-infection or superinfection during COVID disease.

SECONDARY OUTCOMES:
Percentage of coinfected/overinfected patients with severe COVID and the diversity of the pulmonary microbiome. | 24 months
  To observe patterns of lung microbiome diversity in patients with severe COVID that will help us predict the development of coinfection or superinfection in these patients.
Immunologic or cellular patterns in coinfection or superinfection in patients with severe COVID. | 24 months
  To describe immunological or cellular patterns in patients with severe COVID that will help us predict the development of coinfection or superinfection in these patients.

OTHER OUTCOMES:
Type of specimen and conventional cultures for the diagnosis of coinfection or superinfection in patients with severe COVID. | 24 months
  To evaluate three types of respiratory samples by conventional culture for the diagnosis of coinfection or superinfection. This will be compared with the findings of genomic sequencing to be performed to determine the pulmonary microbiome.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad De La Sabana, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
confidentiality agreement